CLINICAL TRIAL: NCT06162897
Title: Implementation of a Triadic Network Case Management Intervention for Individuals Living With or Vulnerable to HIV
Brief Title: Case Management Dyad
Acronym: CM2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB23-0938; 5R01MH131476-02 (NIH)
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-05

CONDITIONS: HIV; Pre-exposure Prophylaxis; Case Management
Keywords: linkage to care; viral suppression; case management; retention in care; financial wellbeing; food security

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (No Intervention): Participants will be offered the current standard of care, Ryan White Non-Medical Case Management. Case management services are need focused and contact is client initiated.
- Dyadic Case Management (Experimental): Participants will receive dyadic case management, specifically they will have two case managers assigned to their case. Case management services will be goal focused and will utilize components from Appreciative Inquiry to orient work to future planning, goals, and financial stability.
  Interventions: Behavioral: Dyadic Case Management

INTERVENTIONS:
Behavioral: Dyadic Case Management — Subjects enrolled in the intervention arm will be offered focused case management centered around goal setting and future orientation. Subjects will be assigned two case managers to support their goals.
  Arms: Dyadic Case Management

SUMMARY:
The overall goal of this study is to test whether dyadic and focused case management will (1) improve financial wellbeing, (2) improve access to food, (3) increase linkage and retention rates for individuals living with HIV or those taking PrEP (PrEP persistence), and (4) increase the proportion of individuals living with HIV who are virally suppressed (viral suppression) when compared to routine Ryan White Non-Medical Case Management.

DETAILED DESCRIPTION:
The purpose of this research is to test the impact of dyadic, focused case management on financial well-being, access to food, linkage to and retention in care outcomes for individuals living with or vulnerable to HIV. The study population is men who have sex with men (MSM) or same-sex attraction, gender-diverse persons, and cis-gender women living with or at increased vulnerability to HIV.

The study team will be testing the hypotheses that dyadic case management that is focused on financial wellness, will have better outcomes for folks living with or vulnerable to HIV. Analyses will be used to assess the efficacy of the intervention as an emerging practice.

ELIGIBILITY:
Gap in HIV or PrEP care access in the past 24 months, defined as a gap greater than 6 months or detectable viral load at least one time in the past 24 months

Self-reported financial or food insecurity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Financial wellbeing | 18 months
  Proportion of subjects who report improved financial wellbeing (e.g. consistent income, ability to pay bills).
Food Security | 18 months
  Proportion of individuals who report improved access to food (e.g. fewer gaps in access to food, reduced concern about access to food).

SECONDARY OUTCOMES:
PrEP Persistence | 18 months
  Proportion of individuals who have engaged in PrEP care regularly (beyond 6 months).
Viral Suppression | 18 months
  Proportion of individuals who have a viral load below 200 copies/mL

CONTACTS AND LOCATIONS:
Overall Officials: John Schneider, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Evans WN, Sullivan JX, Wallskog M. The impact of homelessness prevention programs on homelessness. Science. 2016 Aug 12;353(6300):694-9. doi: 10.1126/science.aag0833. Epub 2016 Aug 11. PMID 27516600
- [Background] Bailey ZD, Krieger N, Agenor M, Graves J, Linos N, Bassett MT. Structural racism and health inequities in the USA: evidence and interventions. Lancet. 2017 Apr 8;389(10077):1453-1463. doi: 10.1016/S0140-6736(17)30569-X. PMID 28402827
- [Background] Singer AW, Weiser SD, McCoy SI. Does Food Insecurity Undermine Adherence to Antiretroviral Therapy? A Systematic Review. AIDS Behav. 2015 Aug;19(8):1510-26. doi: 10.1007/s10461-014-0873-1. PMID 25096896
- [Background] Wheeler DP, Fields SD, Beauchamp G, Chen YQ, Emel LM, Hightow-Weidman L, Hucks-Ortiz C, Kuo I, Lucas J, Magnus M, Mayer KH, Nelson LE, Hendrix CW, Piwowar-Manning E, Shoptaw S, Watkins P, Watson CC, Wilton L. Pre-exposure prophylaxis initiation and adherence among Black men who have sex with men (MSM) in three US cities: results from the HPTN 073 study. J Int AIDS Soc. 2019 Feb;22(2):e25223. doi: 10.1002/jia2.25223. PMID 30768776
- [Background] Lopez JD, Shacham E, Brown T. The Impact of Clinic Policy Attendance and the Ryan White HIV/AIDS Medical Case Management Program on HIV Clinical Outcomes: A Retrospective Longitudinal Study. AIDS Behav. 2020 Apr;24(4):1161-1169. doi: 10.1007/s10461-019-02738-8. PMID 31768689
- [Background] Bouris A, Jaffe K, Eavou R, Liao C, Kuhns L, Voisin D, Schneider JA. Project nGage: Results of a Randomized Controlled Trial of a Dyadic Network Support Intervention to Retain Young Black Men Who Have Sex With Men in HIV Care. AIDS Behav. 2017 Dec;21(12):3618-3629. doi: 10.1007/s10461-017-1954-8. PMID 29079949
- See also: This is the link to the project this study is based on. — https://catholiccharitiesfortworth.org/new-research-on-why-padua-works/